CLINICAL TRIAL: NCT05835505
Title: Detoxification of the Liver in Primary Sclerosing Cholangitis
Brief Title: Detoxification of the Liver In PSC (Dolphin)
Acronym: DOLPHIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000196
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Intervention Model Description: This a crossover study in which everyone will have a period of time on the active medication and a period of time on the placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRS201 Arm (Active Comparator): In Group 1 of the study, subjects will take oral study drug at 1.2g twice daily, PO (2.4g daily) for 4 weeks.
  In Group 2 of the study, subjects will take oral study drug at 2g twice daily, PO (4g daily) for 4 weeks.
  In Group 3 of the study, subjects will take receive a one-time 5g IV dose of the study drug using the FDA-approved IV product followed by the oral study drug at 2g twice daily, PO (4g daily) for 4 weeks.
  In Group 4 of the study, subjects will repeat the previous conditions of the group that proves to be the most effective.
  Interventions: Drug: BRS201
- Placebo Arm (Placebo Comparator): In Group 1 of the study, subjects will take oral placebo at 1.2g twice daily, PO (2.4g daily) for 4 weeks.
  In Group 2 of the study, subjects will take oral placebo at 2g twice daily, PO (4g daily) for 4 weeks.
  In Group 3 of the study, subjects will take receive a one-time 5g IV dose of the study drug using the FDA-approved IV product followed by the oral placebo at 2g twice daily, PO (4g daily) for 4 weeks.
  In Group 4 of the study, subjects will repeat the previous conditions of the group that proves to be the most effective.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRS201 — Groups 1, 2, 3, and 4 will all contain 7 subjects each, with each subject receiving active study drug and placebo in a randomized order; half will receive the placebo first for four weeks followed by active treatment for four weeks, while the other half will receive active treatment for four weeks followed by placebo for four weeks.
  Arms: BRS201 Arm
Drug: Placebo — Groups 1, 2, 3, and 4 will all contain 7 subjects each, with each subject receiving active study drug and placebo in a randomized order; half will receive the placebo first for four weeks followed by active treatment for four weeks, while the other half will receive active treatment for four weeks followed by placebo for four weeks.
  Arms: Placebo Arm

SUMMARY:
This study is a clinical trial being done to investigate the efficacy of drug BRS201 (hydroxocobalamin) as a treatment in patients with primary sclerosing cholangitis. Participation in this study will take 8 weeks long and the study is structured as a cross-over study in which participants will take the study drug for 4 weeks and a placebo drug for 4 weeks in a randomized order in the form of an oral medication. Participation may also involve receiving an IV dose of the medication. The study will require participants to attend 9 study visits, all of which will be remote. Participation will involve taking an oral medication twice daily, tracking the medication in a log, and getting blood drawn and giving a stool sample for a few lab tests throughout the study. For the lab tests, a research nurse will visit the participant in-home for the convenience of the participant.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PSC for at least 6 months based upon cholangiography (ERCP or MRCP) demonstrating intrahepatic and/or extrahepatic biliary strictures, beading or irregularity consistent with PSC.
* ALP > 1.5 times the upper limit of normal (ULN) at screening.
* Subject must either be on a stable dose of ursodeoxycholic acid for > 6 months prior to screening or have been discontinued > 4 weeks prior to screening (enrollment of patients who are on UDCA will be limited to 60% of all enrolled patients).

Exclusion Criteria:

* Anticipated need for liver transplant within one year as determined by Mayo PSC risk score
* Evidence of decompensated liver disease such as variceal bleeding, ascites, or hepatic encephalopathy.
* Evidence of advanced liver disease including MELD score > 10, bilirubin > 3.0, platelet count < 100,000; or INR > 1.4
* Concomitant chronic liver disease including alcohol related liver disease, chronic hepatitis B or C infection, haemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency, non-alcoholic steatohepatitis, autoimmune hepatitis, or primary biliary cholangitis
* Secondary causes of sclerosing cholangitis
* Patients who have a confirmed malignancy or cancer within 5 years except non-melanoma skin cancers
* Treatment with any investigational agents, within two months or 5 half-lives of the investigational product, whichever is longer.
* Active illicit drug or more than moderate alcohol consumption.
* Evidence of bacterial cholangitis within 6 months of enrollment
* In patients with Ulcerative Colitis, or, if Crohn's disease, a need for additional therapy at time of screening.
* Chronic kidney injury (eGFR < 60)
* Pregnancy or lactation
* Uncontrolled hypertension with a systolic BP > 140 and a systolic BP > 90
* Prohibited medications: current use of vitamin C and prednisone
* Patients with a history or risk of cardiovascular conditions, including arrhythmia, long QT syndrome, congestive heart failure, stroke, or coronary artery disease
* Patients with a history of kidney stones
* Congenital or acquired immunodeficiencies
* Other comorbidities including: diabetes mellitus, systemic lupus
* An episode of acute cholangitis within 4 weeks of screening Check eligibility here: https://redcap.link/Checkmyeligibility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Alkaline Phosphatase (ALP) Test Result | 4 weeks
  The primary endpoint for this study is the capacity of BRS201 to normalize alkaline phosphatase levels from baseline (week 0) compared to end of active treatment (4 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Korzenik, MD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States